CLINICAL TRIAL: NCT00260273
Title: Access, Detection and Psychological Treatments
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Ontario Mental Health Foundation (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 107/2004
Record Dates: First submitted 2005-11-28; First posted 2005-12-01 (Estimated); Last update posted 2007-11-08 (Estimated); Status verified 2007-10

CONDITIONS: Psychoses
Keywords: Preventive Therapy; Psychoses; Cognitive Behaviour Therapy
MeSH Terms: conditions — Psychotic Disorders | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): cognitive Behavioural Therapy
  Interventions: Behavioral: Cognitive Behaviour Therapy
- 2 (No Intervention): supportive therapy

INTERVENTIONS:
Behavioral: Cognitive Behaviour Therapy — therapy
  Arms: 1

SUMMARY:
Schizophrenia is one of society's most costly medical conditions and the most severe among psychiatric disorders. One of the most important and exciting new concepts in psychiatry is that detection and intervention very early in the course of schizophrenia offers what may be the field's best practical hope for realizing substantive improvements in the outcome of schizophrenia or schizophrenia spectrum disorders. Thus, we propose a five year program that focuses on three interconnected major research streams: (1) an evaluation of the effectiveness and cost-effectiveness of a model-driven psychological intervention in preventing or delaying the onset of a psychotic illness; (2) a qualitative study of the pathways to mental health at this time of very high risk; and (3) an exploration of the burden to the healthcare and informal caregiver systems associated with this high risk population.

DETAILED DESCRIPTION:
Research Stream 1:

Treatment and Cost Effectiveness The primary aim of Stream 1 is to evaluate the effectiveness of a model-driven psychological intervention, CBT in preventing or delaying the onset of a psychotic illness and to evaluate the effectiveness of CBT in reducing presenting concerns in a sample of help-seeking individuals who have been operationally defined to be at ultra high risk of developing a psychotic illness. CBT will be compared to supportive therapy (ST). We will also examine the cost-effectiveness of a preventive approach. Using a cost-consequence approach, we will examine the cost-effectiveness of CBT versus supportive therapy in addressing psychosis in the "ultra high risk" phase from the perspective of the payer (i.e., the Ministry of Health and Long-Term Care). The hypotheses are:

(i) The time of conversion will be significantly longer for those in the CBT group compared to those in the ST condition.

(ii) The mean level of attenuated psychotic symptoms (SOPS ratings ) will be significantly lower in the CBT group compared to the ST group at the completion of the intervention and at each follow up point.

(iii) Levels of risk factors (measured by CMRS & GHQ2) will be significantly lower in the CBT group compared to the ST group at the completion of the intervention and at each follow up point.

(iv) Levels of depression and anxiety (measured by CDSS, BAS, SPAI2) will be significantly lower in the CBT group compared to the ST group at the completion of the intervention and at each follow up point.

(v) Level of social functioning (measured by SFS2) will be significantly higher in the CBT group compared to the ST group at the termination of the trial and at each follow up point.

(vi) CBT will be more cost-effective than ST.

Research Stream 2:

Pathways to Care The aim of stream 2 is to obtain the in-depth stories of the ways in which those at ultra high risk of developing a psychotic illness come to seek help from mental health services. By mental health services, we include the formal system (specialty mental health & general medical care), lay system (friends, family, self-help), folk system (alternative healers) and human social service system (clergy, teachers, police). These will be sought from both the perspective of youth and from the perspective of their significant others. Multiple case studies using qualitative approaches will focus on the following four elements: 1) social content; 2) social support system, 3) the illness career; and, 4) the treatment system (See Appendix A for detailed components within these elements of the model). These case studies will be employed to further empirically develop theory relating to pathways to mental health care. Theoretical Propositions: The following four theoretical propositions related to pathways to mental health care were formulated based on the Network Episode Model described above. The focus of this stream will be upon the evaluation, refinement and elaboration of these four theoretical propositions. Multiple case study methodology will be employed to further empirically develop theory relating to pathways to mental health care. (i) Family content (e.g., beliefs about and experiences with the medical system), structure (e.g., size, amount of support) and function (e.g., advice, support or coercion) have a critical influence on the pathways to mental health care for youth at ultra high risk for psychosis.(ii) The community and school content, structure and function have a critical influence on the pathways to mental health care for youth at ultra high risk for psychosis.(iii) Problem recognition and the illness experience as perceived by the individual and significant others have a critical influence on the pathways to mental health care for youth at ultra high risk for psychosis.(iv) The content, structure and function (e.g. organizational constraints) of the treatment system have a critical influence on the pathways to mental health care for youth at ultra high risk for psychosis.

Research Stream 3:

Costs of Caring in Psychosis The aim of this third research stream is to explore the burden to the healthcare system and informal caregivers associated with this ultra high risk population. We seek to address three primary questions:

(i) What are the key components affecting the costs of caring for the ultra high risk population? These costs will be considered with respect to both the formal and informal care providers (i.e., service system and family caregivers, respectively).

(ii) What are other psychological costs of caring that informal caregivers face? (i.e. modification in parental work schedules to accommodate their child's needs, impact on other siblings) (iii) Over time, how do the costs of caring change in terms of the economic and psychological costs?

ELIGIBILITY:
Inclusion Criteria:

* Ages 12-30 years·
* Meeting criteria for an "at risk mental state" based on one or more of the 3 Criteria of Prodromal Symptoms (COPS criteria) with severity as determined by ratings on the Scale of Prodromal Symptoms (SOPS) or the criteria for attenuated symptoms of the early prodromal state defined by the presence of at least two of 9 symptoms on the Bonn Scale for the Assessment of Basic Symptoms that have been demonstrated to have the best positive predictive value of developing schizophrenia (Klosterkötter et al., 2001). These criteria for the early prodromal state course are currently used in the multi-site European Prediction of Psychosis Study (EPOS) (Birchwood et al., 2002).

Exclusion Criteria:

* Meets criteria for current or lifetime axis I psychotic disorder.·
* Meets DSM-IV criteria for an Axis 1 disorder where in the judgment of the evaluating clinician the diagnostic prodromal symptoms are clearly caused by the Axis 1 disorder. Note that, except for bipolar and psychotic disorders and a current major depression other DSM-IV disorders will not be exclusionary (e.g. substance abuse or dependence disorder, major depression, anxiety disorders, Axis II Disorders) as long as the disorder does not account for the diagnosis of prodromal symptoms.·
* Use of substances where in the judgment of the evaluating clinician, the diagnostic prodromal symptoms are substance-induced.
* Prior history of treatment with an antipsychotic for the current presenting symptoms or for any previous episode of psychotic symptoms.
* Impaired intellectual functioning (IQ< than 70).
* Past or current history of a clinically significant central nervous system disorder which may confound or contribute to prodromal symptoms.

Ages: 12 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 56 (Actual)
Dates: Start 2004-08; Study Completion 2008-08 (Estimated)

PRIMARY OUTCOMES:
Research Stream 1: Treatment and Cost Effectiveness Primary outcome measure: (i) Time to conversion. | 18 months
Research Stream 2: Pathways to Care Primary outcome measure: Pathway to care interview | 18 months
Research Stream 3: Costs of Caring in Psychosis Primary outcome measure: (i) Time to conversion, (ii) costs of formal and informal care giving. | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Jean Addington, PhD, Principal Investigator — Centre for Addiction and Mental Health/ University of Toronto
Locations (1):
- Centre for Addiction and Mental Health, Toronto, Ontario, Canada